CLINICAL TRIAL: NCT00569439
Title: A Randomized Controlled Trial Comparing Normal Saline With and Without Dextrose on the Course of Labor in Nulliparas
Brief Title: A Study on the Effects of Dextrose Solutions on the Course of Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MemorialCare (Other)
Responsible Party: Kenneth Chan, Memorial Care
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 035-00
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2006-06

CONDITIONS: Labor
Keywords: Labor; Carbohydrate; Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- D5 (Experimental): 5% Dextrose Solution in Normal Saline
  Interventions: Drug: D5NS
- D10 (Experimental)
  Interventions: Drug: D10NS
- NS (Placebo Comparator)
  Interventions: Drug: NS

INTERVENTIONS:
Drug: D5NS — 5% Dextrose in Normal Saline (6.25 gr/hr) at 125 cc/hr
  Arms: D5
Drug: D10NS — 10% Dextrose Solution (12.5 gr/h) in Normal Saline at 125 cc/hr
  Arms: D10
Drug: NS — Normal Saline solution at 125 cc/hr
  Arms: NS

SUMMARY:
The purpose is to determine in term nulliparas with singletons that present in active labor (3-5 cm) or with ruptured membranes whether the administration of dextrose solutions to normal saline improves or expedites the course of labor. The researchers' hypothesis is that the addition of a carbohydrate substrate will shorten the length of labor and facilitate a vaginal delivery.

DETAILED DESCRIPTION:
Factors that affect the course of labor have been studied extensively. Surprisingly, there is little data on the effect that different types and rates of intravenous (IV) fluids have during labor. Exercise physiologists have shown that increased fluid intake and carbohydrate replacement improve skeletal muscle performance in prolonged exercise. In a 1992 randomized, controlled study comparing IV fluid rates, Garite et al. showed a lower frequency of prolonged labor, and possibly a decreased need for oxytocin, with higher IV fluid rates in labor. Inadequate hydration may contribute to dysfunctional labor and possibly an increased rate of cesarean section.

We propose that inadequate carbohydrate replacement in labor may also contribute to prolongation of labor and increased need for operative delivery. Glucose is the main energy supply for the pregnant uterus. Physiological requirements for glucose during labor are approximately 10 grams per hour. Adequate supplies of glucose are needed to maintain exercise tolerance and muscle efficiency, which are important factors in the progress of labor. Dysfunctional labor or dystocia, which is the leading indication for primary cesarean delivery, is caused by uterine forces insufficiently strong or inappropriately coordinated to efface and dilate the cervix. Dystocia can also be a result of inadequate voluntary muscle effort in the second stage of labor. It contributes to increased risk for chorioamnionitis, which is a leading cause of maternal and fetal morbidity and mortality. Supplying carbohydrate fuel for working uterine and skeletal muscle may improve progress in labor and, therefore, diminish risk for chorioamnionitis and need for cesarean delivery.

ELIGIBILITY:
* Primiparous
* Singleton gestation
* Vertex presentation
* Spontaneous active labor with or without pitocin augmentation
* Gestational age > 36 weeks
* Cervical dilation 3 to 5 cm with or without ruptured membranes

Exclusion Criteria:

* Multiparous
* Pregestational or gestational diabetes mellitus
* Preeclampsia at admission
* Previous cesarean section
* Non-vertex presentation
* Multiple gestation
* Chorioamnionitis at admission
* Intrauterine growth restriction (< 10th percentile)
* Patients admitted for induction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2000-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Carbohydrate solutions can decrease the total duration of labor by 20% (from 560 minutes to 450 minutes) | Prospective

SECONDARY OUTCOMES:
Carbohydrate solutions can decrease the incidence of prolonged labor (> 12 hours | Prospective
Carbohydrate solutions can decrease the incidence of chorioamnionitis during labor | Prospective
Carbohydrate solutions can decrease the need for oxytocin (a contraction stimulant) augmentation of labor | Prospective
Carbohydrate solutions can decrease the frequency of cesarean sections for prolonged labor | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chan, M.D., Principal Investigator — Memorial Care; Sherri Jenkins, M.D., Principal Investigator — University of Alabama at Birmingham; Thomas J. Garite, M.D., Principal Investigator — University of California, Irvine